CLINICAL TRIAL: NCT04567914
Title: Ultrasonographic Evaluation of Abdominal Muscle Thickness Symmetry and Correlation With Pulmonary Function Test in Adolescent Idiopathic Scoliosis
Brief Title: Ultrasonographic Evaluation of Abdominal Muscle Thickness Symmetry and Correlation With Pulmonary Function
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: IstPMRTRH-SCO1
Record Dates: First submitted 2020-09-24; First posted 2020-09-29 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Muscle Physiology; Adolescent Idiopathic Scoliosis
Keywords: Abdominal muscle; Cobb angle; Imbalance; Spirometry; Ultrasonography
MeSH Terms: interventions — Ultrasonography; Spirometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adolescent idiopathic scoliosis: Ultrasonographic measurements were performed of bilaterally abdominal muscle thickness of AIS patients diagnosed by a specialist. Spirometry evaluation was performed by the investigator
  Interventions: Diagnostic Test: Bilaterally abdominal muscle thickness with ultrasonography
- Adolescent healthy individuals: Healthy adolescents aged 10-18 were selected. Ultrasonographic measurements were performed of bilaterally abdominal muscle thickness. Spirometry evaluation was performed by the investigator.
  Interventions: Diagnostic Test: Bilaterally abdominal muscle thickness with ultrasonography

INTERVENTIONS:
Diagnostic Test: Bilaterally abdominal muscle thickness with ultrasonography — AIS group was evaluated for localization of curvature and degree of curvature. Ultrasonographic measurements were performed of bilaterally abdominal muscle thickness in the supine and standing positions in both groups. Spirometry evaluation was performed in both groups
  Other Names: Spirometry

SUMMARY:
We aimed in this study:

1. To compare the ultrasonographic measurements of the abdominal muscles thickness symmetry in patients with adolescent idiopathic scoliosis (AIS) and adolescent healthy individuals
2. To investigate the effect of measured thickness and symmetry on pulmonary function test.

DETAILED DESCRIPTION:
This cross-sectional,case-control clinical study included 40 patients diagnosed with AIS and 40 age and gender -matched healthy individuals. AIS group was evaluated for localization of curvature and degree of curvature. Ultrasonographic measurements and were performed of bilaterally abdominal muscle thickness in both groups. Spirometry evaluation was performed in both groups. Intragroup and intergroup data were compared.

ELIGIBILITY:
Inclusion Criteria:

* Cobb angle over 10 degrees in radiological evaluation
* Between the ages of 10-18 and diagnosed with AIS by a specialist physiatrist

Exclusion Criteria:

* History of previous spinal surgery
* Patients using brace
* Those with any diagnosis of scoliosis other than AIS
* Those with a history of neuromuscular disease
* Previous spinal surgery
* Patients with neurological deficits on examination
* Patients with acute or chronic lung pathology
* Patients with abdominal surgery or injury
* Double curve or multiple curve
* Patients with concomitant chronic diseases
* The child's legal guardian does not allow it to take the tests

The control group:

* 10-18 volunteer adolescents without any health problems,
* In clinical evaluation: Healthy adolescents (without any asymmetric findings on three-way inspection, Adam's forward bend test and scoliometer) were included.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 10-18 years old patient with AIS diagnosis 10-18 years old healthy adolescent volunteer
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Abdominal Muscle Thickness Symmetry | during evaluation, an average of 45 minutes
  bilateral ultrasonographic millimetric measurement

SECONDARY OUTCOMES:
Spirometry | during evaluation, an average of 30 minutes
  Forced expiratory volume 1 (FEV1), Forced vital capacity (FVC), FEV1/FVC, Peak expiratory flow (PEF)
Cobb angle | during evaluation, an average of 30 minutes
  Measurements were made on orthoroentgenogram, Grouped as Cobb angle <20 and Cobb angle ≥20

CONTACTS AND LOCATIONS:
Overall Officials: Muhsin DORAN, MD, Principal Investigator — Istanbul Physical Medicine Rehabilitation Training and Research Hospital; Kadriye Öneş, Assoc Prof, Study Chair — Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teyhen DS, Gill NW, Whittaker JL, Henry SM, Hides JA, Hodges P. Rehabilitative ultrasound imaging of the abdominal muscles. J Orthop Sports Phys Ther. 2007 Aug;37(8):450-66. doi: 10.2519/jospt.2007.2558. PMID 17877281
- [Background] Newton PO, Faro FD, Gollogly S, Betz RR, Lenke LG, Lowe TG. Results of preoperative pulmonary function testing of adolescents with idiopathic scoliosis. A study of six hundred and thirty-one patients. J Bone Joint Surg Am. 2005 Sep;87(9):1937-46. doi: 10.2106/JBJS.D.02209. PMID 16140807
- [Result] Linek P. Body Mass Normalization for Lateral Abdominal Muscle Thickness Measurements in Adolescent Athletes. J Ultrasound Med. 2017 Sep;36(9):1851-1857. doi: 10.1002/jum.14218. Epub 2017 May 15. PMID 28503815
- [Result] Yang HS, Yoo JW, Lee BA, Choi CK, You JH. Inter-tester and intra-tester reliability of ultrasound imaging measurements of abdominal muscles in adolescents with and without idiopathic scoliosis: a case-controlled study. Biomed Mater Eng. 2014;24(1):453-8. doi: 10.3233/BME-130830. PMID 24211927
- [Result] Dreimann M, Hoffmann M, Kossow K, Hitzl W, Meier O, Koller H. Scoliosis and chest cage deformity measures predicting impairments in pulmonary function: a cross-sectional study of 492 patients with scoliosis to improve the early identification of patients at risk. Spine (Phila Pa 1976). 2014 Nov 15;39(24):2024-33. doi: 10.1097/BRS.0000000000000601. PMID 25202929